CLINICAL TRIAL: NCT07264244
Title: Delirium Incidence and Indwelling Urinary CathEterization After Acute Stroke
Acronym: DICES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: all participants recruited
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 144/2021BO1
Record Dates: First submitted 2021-04-06; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2021-03

CONDITIONS: Post-Stroke Delirium

STUDY DESIGN:
Intervention Model Description: randomised open label trial
Who Masked: Outcomes Assessor
Masking Description: outcome assessor is masked for intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual care (IUC) (No Intervention)
- condom catheter (Active Comparator)
  Interventions: Device: condom catheter

INTERVENTIONS:
Device: condom catheter — The subjects will be randomly assigned to one of two groups. The subjects in the control group will receive as part of our ongoing clinical routine an IUC at the time of admission. For IUC a well established standard operating procedure in our clinic will be followed (https://vswroxtra01.ukt.ad.local/Roxtra/index.aspx: Legen eines transurethralen Blasenkatheters (BLK). The intervention group will be provided a condom catheter. If necessary, the ladder will be assisted with a urine bottle or a toilet chair
  Arms: condom catheter

SUMMARY:
The main goal of this study is to identify indwelling urinary catheterization (IUC) as a predictive factor of the development of delirium in male acute stroke patients.

DETAILED DESCRIPTION:
The main goal of this study is to identify indwelling urinary catheterization (IUC) as a predictive factor of the development of delirium in male acute stroke patients. With a prospective randomized-controlled interventional study design it aims to provide reliable evidence to effectively reduce delirium as well as secondary complications after IUC in critically ill patients. Until now, male, severely affected acute stroke patients regularly receive IUC for recanalization therapy or to balance fluid intake. Complications might be urinary infections, agitation and accidental removal by the patient himself with urinary bleeding.

We ought to investigate if early removal of the IUC after recanalization therapy and replacement with either a condom catheter or a diaper might reduce complications after catheterization and hereby reduce delirium.

As a secondary outcome we would like to explore other options besides indwelling urinary catheterization for balancing the fluid in- and output.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria

* Male gender
* Age ≥ 70 years
* Treated with recanalization therapy and therefore receiving an IUC
* Patient is able to provide written informed consent. If patient is aphasic and not in a position to provide written informed consent after the stroke, a relative or a legal guardian can provide information of the presumed will of the patient.

Inclusion of this patient is possible if the patient will give basic informed consent as soon as he is able to and after a maximum of seven days after enrollment.

As delirium is associated with stroke severity it is necessary to include these patients, otherwise the incidence of delirium will be too low.

Exclusion Criteria:

* Delirium at admission
* Need for mechanical ventilation > 48h
* Presence of an IUC before admission

Min Age: 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — male
Enrollment: 50 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Delirium | 10 days after admission
  The primary outcome will be the development of delirium within 10 days after admission.
  Secondary outcomes will be
  * Length of stay on NICU / stroke unit
  * Development of UTI
  * Development of neurological bladder dysfunction
  * Pleura effusions and/or ankle edema

CONTACTS AND LOCATIONS:
Overall Officials: Annerose Mengel, MD, Principal Investigator — Universitätsklnikum Tübingen
Locations (1):
- University Medicine Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided